CLINICAL TRIAL: NCT05179356
Title: Effects of DAPAgliflozin on Cardiopulmonary Exercise Capacity and Hemodynamics in Pulmonary Arterial Hypertension: A Double Blind Randomized Trial. (DAPAH-trial)
Brief Title: Dapagliflozin in Pulmonary Arterial Hypertension
Acronym: DAPAH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mads Ersbøll (Other)
Responsible Party: Sponsor-Investigator, Mads Ersbøll, Medical doctor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAPAH16122021
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Arterial Hypertension; Chronic Thromboembolic Pulmonary Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin 10 mg once daily (Active Comparator): Dapagliflozin 10 mg (Farxiga 10 mg) given once daily for three months
  Interventions: Drug: Dapagliflozin 10 MG [Farxiga]
- Matching placebo (Placebo Comparator): Placebo given once daily for three months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10 MG [Farxiga] — Dapagliflozin 10 mg given once daily for three months
  Arms: Dapagliflozin 10 mg once daily
Drug: Placebo — Matching placebo
  Arms: Matching placebo

SUMMARY:
The purpose of this study is to investigate the effects of dapagliflozin on exercise capacity and hemodynamics in patients with pulmonary arterial hypertension

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effects of oral dapagliflozin (Forxiga®) treatment versus placebo in clinically stable patients with pulmonary arterial hypertension or CTEPH on background vasodilator combination therapy on cardio-pulmonary exercise capacity, pulmonary vascular hemodynamics, RV function and metabolomic profile of the pulmonary vascular endothelium.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of PAH group 4 or group 1 in any of the following subtypes:

  * Idiopathic PAH (iPAH)
  * Heritable PAH (hPAH)
  * Connective tissue disease associated PAH (aPAH)
  * Associated with congenital heart disease (aPAH)
  * In case of PH in group 4, no further invasive treatment including pulmonary endarterectomy or pulmonary balloon angioplasty must be planned at time of inclusion.
* Symptomatic PAH in WHO functional class II-III as assessed by the screening clinician.
* Clinically stable patients on pulmonary vasodilator treatment with PDE5i, ERA, PA/IPA alone or in combination without considerations from the treating physician team towards treatment escalation and a treatment duration of at least four weeks. Clinical stability defined as stable symptoms without progression as assessed by treating clinician and without the need for unplanned hospital admissions due to worsening PAH within three months of screening.
* Fertile women (< 50 years of age) must use safe contraceptives (Intra uterine device or hormonal contraception) for the duration of the study and have a negative pregnancy test
* Able to understand the written patient information in Danish and give informed consent.
* Age ≥ 18 years
* Ability to perform cardio pulmonary exercise test

Exclusion Criteria:

* Known allergy to the study medication
* Treatment with an SGLT2i within 6 months prior to baseline
* Type 1 or type 2 diabetes
* Impaired renal function with an eGFR < 30 mL/min/m2 within four weeks of screening
* Severe liver dysfunction (Child-Pugh class c)
* Listed for lung transplantation at the time of screening
* Planned initiation of iv prostacyclin therapy/ IPA or current dose escalation planned
* Planned pulmonary endarterectomy or pulmonary balloon angioplasty.
* LVEF < 50%
* Diagnosis of PAH group 2, 3 or 5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-01-13 (Actual); Study Completion 2026-01-13 (Actual)

PRIMARY OUTCOMES:
Change in VO2 max from baseline to follow up | 3 months

SECONDARY OUTCOMES:
Change in 6 minutes walking distance | 3 months
Change in VE/VCO2 | 3 months
Change in pulmonary vascular resistance | 3 months
Change in mean pulmonary artery pressure | 3 months
Change in Cardiac index | 3 months
Change in central venous pressure | 3 months
Change in transpulmonary gradient | 3 months
Change in pulmonary arterial compliance | 3 months
Change in right ventricular size on 3D echocardiography | 3 months
Change in right ventricular free wall strain | 3 months
Change in right ventricular free wall strain-work (free wall strain/ pulmonary artery pressure) | 3 months
Change in NTproBNP | 3 months
Change in EQ-5D-5L questionnaire | 3 months
Change in metabolomic pattern on central venous blood | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No